CLINICAL TRIAL: NCT02819076
Title: EVENDOL Scale Validation for at Term New-born
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EVENDOL
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Painless Children: 30 children
  Interventions: Other: pain scale
- Painful Children: 70 children
  Interventions: Other: pain scale

INTERVENTIONS:
Other: pain scale

SUMMARY:
Maternity and neonatology, caregivers are regularly confronted with the pain of the newborn, especially after a birth injury, but it is sometimes difficult ti define.

There is not, to our knowledge, any prevalence study of pain in newborn motherhood. The data available are those of the perinatal survey 2010, with the number of operative vaginal deliveries (5.3% of suction, forceps 3.9%, 2.9% spatulas) and the number of extractions the seat (4.7%). These delivery modes can be purveyors of pain.

At St. Joseph's Hospital, there were in 2013: 259 instrumental deliveries and 90 extractions by headquarters. Fifty five paracetamol bottles were consumed in the layer sequence in 2013, and 15 in the delivery room. But this consumption is a poor reflection of the pain because treatment could be given pain-authenticated (measured with the EDIN scale), and because a bottle is discarded one month after opening.

The scales measuring pain used in the new-born at term based on the assessment of change in behavior; two specific scores of the newborn are used in France: Pain and Discomfort Scale Newborn (EDIN) for prolonged pain and Acute Pain scale Newborn (DAN) for acute pain related to health care.

The EVENDOL scale (Child Pain Evaluation) has been validated for pediatric emergencies in children 0-7 years, as well as pre-hospital, to measure the intensity of pain whether acute or prolonged (8 ). It is easy and fast to use. validation cohorts included a significant proportion of newborns. This scale appears suitable for evaluation of the newborn to term maternity

DETAILED DESCRIPTION:
Objectives:

Principal: validation of the instrument "EVENDOL" in the new-born at term.

Secondary:

* EVENDOL is equivalent to EDIN to diagnose the pain of the newborn at term.
* While being faster and easier to dimension.
* EVENDOL preferred by caregivers

Methodology and conduct of the study:

DESIGN: Study of practical evaluation of observational, prospective, multicenter.

Places of study: maternity of Saint Joseph Hospital, and Kremlin Bicetre. A feasibility study is underway, it was started in neonatology Antoine Béclère. Time study: 12 to 18 months Required subjects: 100 patients (1/3 painless children, 2/3 of painful children).

ELIGIBILITY:
Inclusion Criteria:

* New born at term (≥ 37 weeks)
* Suspects or without pain
* From 0 to 28 days of life,
* Able to be studied and monitored by the researcher.

Exclusion Criteria:

* Prematurity: newborn <37 SA
* Children in intensive care or intensive care unit
* Children in vital distress
* Major malformation syndrome
* Non-Francophone Parents

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This scale appears suitable for evaluation of the newborn at term pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Assessment of change in EVENDOL scale | 0 minute, 45 minutes then 90 minutes
Assessment of change in EDIN (Pain and Discomfort Scale Newborn) scale | 0 minute, 45 minutes then 90 minutes
Assessment of change in NFCS (Neonatal Facial Coding System) scale | 0 minute, 45 minutes then 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Walter Elisabeth, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Hôpital Armand Trousseau, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

REFERENCES:
- [Derived] Calamy L, Fournier-Charriere E, Martret P, Cimerman P, Boithias C, Debillon T, Carbajal R, Falissard B, Walter-Nicolet E. The EVENDOL Pain Scale Validation for Acute Non-Procedural Neonatal Pain in Term Neonates: Reliability and Validity in Maternity Wards. Paediatr Neonatal Pain. 2025 Jun 6;7(2):e70008. doi: 10.1002/pne2.70008. eCollection 2025 Jun. PMID 40487028